CLINICAL TRIAL: NCT00508404
Title: A Single Arm Multicentre Phase II Study of Panitumumab in Combination With Irinotecan/5-fluorouracil/Leucovorin in Patients With Metastatic Colorectal Cancer
Brief Title: Panitumumab Plus FOLFIRI in First-line Treatment of Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060314; EUDRACT Number 2006-006739-36
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Results first posted 2016-01-26 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab plus FOLFIRI (Experimental): Participants received 6 mg/kg panitumumab intravenously (IV) once every 14 days in combination with FOLFIRI chemotherapy regimen consisting of irinotecan, infusional 5-fluorouracil, and leucovorin, until diagnosed with radiographic disease progression.
  Interventions: Drug: Panitumumab; Drug: FOLFIRI

INTERVENTIONS:
Drug: Panitumumab — Administered by intravenous infusion
  Other Names: Vectibix
Drug: FOLFIRI — FOLFIRI chemotherapy was initiated on Day 1 of each treatment cycle at the following starting doses: irinotecan 180 mg/m², leucovorin 400 mg/m², 5-fluorouracil bolus 400 mg/m², 5-fluorouracil infusion 2400 mg/m².

SUMMARY:
To estimate the effect of KRAS mutation status (Wild-type versus Mutant) on objective response rate and other measures of efficacy for patients treated with panitumumab in combination with a chemotherapy regimen of irinotecan, 5-fluorouracil, and leucovorin (FOLFIRI) as first-line therapy for metastatic colorectal cancer (mCRC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with histologically- or cytologically-confirmed metastatic adenocarcinoma of the colon and/or rectum.
* Measurable disease according to modified RECIST guidelines.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Paraffin-embedded tissue or unstained tumour slides from primary or metastatic tumour available for central lab analysis.
* Adequate haematologic, renal, hepatic and metabolic function.

Exclusion Criteria:

* Central nervous system metastases.
* Prior systemic therapy for the treatment of metastatic colorectal carcinoma with the exception of adjuvant fluoropyrimidine-based chemotherapy given at least six months prior to initiating study treatment.
* Prior anti-epidermal growth factor receptor (EGFr) antibody therapy (e.g. cetuximab) or treatment with small molecule EGFr tyrosine kinase inhibitors (e.g. erlotinib).
* Prior radiotherapy within 14 days prior to screening, and for which all signs of early radiological toxicity have not abated.
* Significant cardiovascular disease including unstable angina or myocardial infarction within six months before initiating study treatment or a history of ventricular arrhythmia.
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline chest computed tomography (CT scan.
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhoea (defined as > 4 loose stools per day).
* History of Gilbert's syndrome or dihydropyrimidine deficiency.
* Known positive test for human immunodeficiency virus infection, hepatitis C virus, chronic active hepatitis B infection.
* Any investigational agent within 30 days before initiation of study treatment.
* Must not have had a major surgical procedure within 28 days prior to initiation of study treatment.
* Subject who is pregnant or breast-feeding.
* Woman or man of childbearing potential not consenting to use adequate contraceptive precautions during the course of the study and for six months after the last study drug administration for women, and one month for men.

  * Other protocol specified criteria and specific details may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2007-05-09 (Actual); Primary Completion 2009-06-01 (Actual); Study Completion 2012-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Kohne CH, Hofheinz R, Mineur L, Letocha H, Greil R, Thaler J, Fernebro E, Gamelin E, Decosta L, Karthaus M. First-line panitumumab plus irinotecan/5-fluorouracil/leucovorin treatment in patients with metastatic colorectal cancer. J Cancer Res Clin Oncol. 2012 Jan;138(1):65-72. doi: 10.1007/s00432-011-1061-6. Epub 2011 Sep 30. PMID 21960318
- [Background] Thaler J, Karthaus M, Mineur L, Greil R, Letocha H, Hofheinz R, Fernebro E, Gamelin E, Banos A, Kohne CH. Skin toxicity and quality of life in patients with metastatic colorectal cancer during first-line panitumumab plus FOLFIRI treatment in a single-arm phase II study. BMC Cancer. 2012 Sep 29;12:438. doi: 10.1186/1471-2407-12-438. PMID 23020584
- [Derived] Taieb J, Geissler M, Rivera F, Karthaus M, Wilson R, Loupakis F, Price T, Tracy M, Burdon P, Peeters M. Relationship Between Tumor Response and Tumor-Related Symptoms in RAS Wild-Type Metastatic Colorectal Cancer: Retrospective Analyses From 3 Panitumumab Trials. Clin Colorectal Cancer. 2019 Dec;18(4):245-256.e5. doi: 10.1016/j.clcc.2019.07.009. Epub 2019 Jul 29. PMID 31515083
- [Derived] Kohne CH, Karthaus M, Mineur L, Thaler J, Van den Eynde M, Gallego J, Koukakis R, Berkhout M, Hofheinz RD. Impact of Primary Tumour Location and Early Tumour Shrinkage on Outcomes in Patients with RAS Wild-Type Metastatic Colorectal Cancer Following First-Line FOLFIRI Plus Panitumumab. Drugs R D. 2019 Sep;19(3):267-275. doi: 10.1007/s40268-019-0278-8. PMID 31300973
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 169 patients were screened, of whom 154 were enrolled into this study at 36 study centers in Austria, Belgium, France, Germany, and Sweden from 9 May 2007 through 18 June 2008.
  Results are reported through the primary analysis data cut-off date of 18 June 2009 (12 months after the last patient was enrolled).
Pre-assignment Details: Participants received a FOLFIRI regimen in combination with panitumumab once every 14 days until diagnosed with radiographic disease progression, at which time the participant was withdrawn from the treatment phase. Participants were to complete a safety follow-up visit 8 weeks after the treatment phase.
Period: Overall Study
Arm/Group | Panitumumab Plus FOLFIRI
Started | 154
Completed | 112 (Completion of safety follow-up visit conducted 8 weeks after last dose)
Not Completed | 42
Not completed — Ongoing at Data Cut-off | 12
Not completed — Adverse Event | 2
Not completed — Death | 16
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 3
Not completed — Protocol-specified Criteria | 2
Not completed — Lost to Follow-up | 2
Not completed — Other - Not Specified | 3

BASELINE CHARACTERISTICS:
Arm/Group | Panitumumab Plus FOLFIRI
Number analyzed (Participants) | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 105
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 2
  Hispanic or Latino | 1
  Japanese | 1
  White or Caucasian | 150
Kirsten Rat Sarcoma-2 Virus (KRAS) Mutation Status [Number; unit: participants]
  Wild-type KRAS | 86
  Mutant KRAS | 59
  Unevaluable KRAS | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate is defined as the percentage of participants with a best response of complete response or partial response. Disease assessments are based on investigator review of scans using modified Response Evaluation Criteria in Solid Tumors (RECIST) V1.0 criteria. A complete or partial response was confirmed no less than 4-weeks after the criteria for response were first met. Participants with no post-baseline assessment were considered non-responders.
  Complete Response (CR): disappearance of all target and non-target lesions and no new lesions.
  Partial Response (PR): At least a 30% decrease in the size of target lesions with no progression of non-target lesions and no new lesions, or, the disappearance of all target lesions but persistence of 1 or more non-target lesions not qualifying for either CR or progressive disease (PD) and no new lesions.
Time Frame: Tumor response was assessed at Week 8 and every 8 weeks to Week 48 and 3 monthly thereafter until disease progression; median follow-up time was 34 weeks
Population: KRAS Tumor Response Analysis Set (all participants who provided informed consent, enrolled, received at least 1 dose of panitumumab, had evaluable KRAS status data, and with at least 1 unidimensionally measurable lesion per modified RECIST by the local investigator)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Wild-type KRAS: Participants with wild-type KRAS received 6 mg/kg panitumumab intravenously (IV) once every 14 days in combination with FOLFIRI chemotherapy regimen consisting of irinotecan, infusional 5-fluorouracil, and leucovorin, until diagnosed with radiographic disease progression.
- Mutant KRAS: Participants with mutant KRAS received 6 mg/kg panitumumab intravenously (IV) once every 14 days in combination with FOLFIRI chemotherapy regimen consisting of irinotecan, infusional 5-fluorouracil, and leucovorin, until diagnosed with radiographic disease progression.
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 85 | 58
percentage of participants | 56.47 [45.28 to 67.20] | 37.93 [25.51 to 51.63]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.02 to 4.45] — The odds ratio is defined as the odds of having an objective response in the KRAS Wild-type group relative to the odds in the KRAS Mutant group

2. Secondary Outcome: Objective Response by 17 Weeks
Description: The percentage of participants with a best response of complete response or partial response by Week 17. Disease assessments are based on investigator review of scans using modified RECIST V1.0 criteria. A complete or partial response was confirmed no less than 4-weeks after the criteria for response were first met. Participants with no post-baseline assessment were considered non-responders.
Time Frame: Up to Week 17
Population: KRAS Tumor Response Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 85 | 58
percentage of participants | 49.41 [38.39 to 60.48] | 34.48 [22.49 to 48.12]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Odds Ratio (OR) = 1.86, 95% CI 2-sided [0.88 to 3.93] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Disease Control Rate
Description: The percentage of participants whose best response was either a complete or partial response or stable disease, based on modified RECIST v1.0 criteria as assessed by the Investigator.
  Stable diease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD of target lesions and no progression of existing non-target lesions and no new lesions, or, the persistence of 1 or more non-target lesions not qualifying for either CR or PD if no target lesions were identified at Baseline.
Time Frame: as for outcome 1
Population: KRAS Tumor Response Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 85 | 58
percentage of participants | 90.59 [82.29 to 95.85] | 89.66 [78.83 to 96.11]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.30 to 3.89] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Duration of Response
Description: Duration of response was calculated only for those participants who had a confirmed complete or partial response, and is defined as the time from first confirmed response to first observed progression. For participants who responded and did not progress by the analysis data cut-off date, duration of response was censored at their last evaluable disease assessment date. Duration of response was analyzed using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: KRAS Tumor Response Analysis Set with an objective response (CR or PR)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 48 | 22
months | 13.0 [9.3 to 13.0] | 7.4 [5.4 to 8.8]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.283, 95% CI 2-sided [0.130 to 0.614] — Hazard ratio is presented as Wild-type KRAS:Mutant KRAS. A value < 1.0 indicates a lower average event rate and longer time to event for Wild-type KRAS relative to Mutant KRAS

5. Secondary Outcome: Time to Initial Objective Response
Description: Time to response is the time from the date of enrollment to the date of first confirmed complete or partial response. Participants with a best response of stable disease at the analysis data cut-off date were censored at their last assessment of SD and participants with all other categories of best response were censored at the maximum observed time to a first confirmed response among all responders. Time to initial objective response was analyzed using Kaplan-Meier methods.
Time Frame: as for outcome 1
Population: KRAS Tumor Response Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 85 | 58
months | 3.8 [3.4 to NA] — Could not be estimated due to the low number of events. | NA [5.5 to NA] — Could not be estimated due to the low number of events.
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Hazard Ratio (HR) = 1.642, 95% CI 2-sided [0.990 to 2.721] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is the time from the date of enrollment to the date of first observed progression or death, whichever comes first. Participants who were alive and did not progress by the analysis data cut-off date were censored at the last evaluable disease assessment date. Progression-free survival was analyzed using Kaplan-Meier methods.
Time Frame: From enrollment until the data cut-off date of 18 June 2009; median follow-up time was 34 weeks.
Population: Primary Analysis Set (all participants who provided informed consent, enrolled, received at least 1 dose of panitumumab, and had evaluable KRAS status data)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 86 | 59
months | 8.9 [7.6 to 14.3] | 7.2 [5.6 to 7.8]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.464, 95% CI 2-sided [0.306 to 0.703] — Hazard ratio presented as Wild-type KRAS:Mutant KRAS. A value < 1.0 indicates a lower average event rate and longer time to event for Wild-type KRAS relative to Mutant KRAS

7. Secondary Outcome: Time to Disease Progression
Description: Time to progression is the time from the enrollment date to the date of first observed progression. For participants who had not progressed by the analysis data cutoff date, time to progressive disease was censored at their last evaluable disease assessment date. Time to disease progression was analyzed using Kaplan-Meier methods.
Time Frame: From enrollment until the data cut-off date of 18 June 2009; median follow-up time was 34 weeks.
Population: Primary Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 86 | 59
months | 11.2 [7.6 to 14.8] | 7.3 [5.7 to 8.9]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.395, 95% CI 2-sided [0.252 to 0.618] — [estimate comment as in outcome 4, analysis 1]

8. Secondary Outcome: Duration of Stable Disease
Description: Duration of stable disease was calculated only for participants with a best response of stable disease and is defined as the time from enrollment to first observed PD. For participants who did not progress by the analysis data cut-off date, duration of SD was censored at their last evaluable disease assessment date. Duration of stable disease was estimated using Kaplan-Meier methods.
Time Frame: as for outcome 1
Population: KRAS Tumor Response Analysis Set with a best response of SD
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 29 | 30
months | 5.9 [5.8 to 7.6] | 6.1 [4.8 to 7.4]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.756, 95% CI 2-sided [0.400 to 1.430] — [estimate comment as in outcome 4, analysis 1]

9. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as the time from enrollment to the date the decision was made to end the treatment phase for any reason. For participants who remained in the treatment phase at the analysis data cut-off date, time to treatment failure was censored at the date of their last on-study assessment. Time to treatment failure was analyzed using Kaplan-Meier methods.
Time Frame: From enrollment until the data cut-off date of 18 June 2009; median follow-up time was 34 weeks.
Population: Primary Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 86 | 59
months | 6.9 [6.2 to 7.6] | 5.8 [5.3 to 6.8]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Hazard Ratio (HR) = 0.710, 95% CI 2-sided [0.503 to 1.002] — [estimate comment as in outcome 4, analysis 1]

10. Secondary Outcome: Time to Disease Relapse Following Surgical Intervention
Description: Calculated only for those participants who underwent surgical intervention, and defined as the time from the date of first post-intervention radiographic disease assessment to the date of first observed PD. Participants with no post-intervention disease assessment had their time to relapse set to zero and censored in the analysis. Participants that had evidence of progression / recurrence at their first post-intervention disease assessment had a time to relapse of zero. For participants who had not progressed by the analysis data cut-off date, time to relapse was censored at the date of their last evaluable disease assessment. Time to relapse was analyzed using Kaplan-Meier metjhods.
Time Frame: From enrollment until the data cut-off date of 18 June 2009; median follow-up time was 34 weeks.
Population: Primary Analysis Set participants who underwent surgery
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 13 | 4
months | NA [NA to NA] — Could not be estimated due to the low number of events. | NA [NA to NA] — Could not be estimated due to the low number of events.

11. Secondary Outcome: Resection Rate
Description: The percentage of participants who underwent a surgical procedure that resulted in partial reduction or complete eradication of all metastatic disease.
Time Frame: From enrollment until the data cut-off date of 18 June 2009; median follow-up time was 34 weeks.
Population: Primary Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Wild-type KRAS | Mutant KRAS
Number analyzed (Participants) | 86 | 59
percentage of participants | 15.12 [8.30 to 24.46] | 6.78 [1.88 to 16.46]
Statistical Analysis 1: Comparison: Wild-type KRAS vs Mutant KRAS; Test type: Superiority or Other; Difference in rates = 8.34, 95% CI 2-sided [-4.01 to 19.08]

ADVERSE EVENTS:
Time Frame: The time frame for adverse event reporting is from the first dose date to 30 days since the last dose date. The median time frame is 6.6 months.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Panitumumab Plus FOLFIRI
Serious Adverse Events (participants affected / at risk) | 84/154
Other Adverse Events (participants affected / at risk) | 154/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus FOLFIRI (N=154)
ANAEMIA (Blood and lymphatic system disorders) | 2
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 6
MYOPERICARDITIS (Cardiac disorders) | 1
CONJUNCTIVITIS (Eye disorders) | 1
OCULAR TOXICITY (Eye disorders) | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 4
ANAL FISSURE (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 21
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 1
FAECALOMA (Gastrointestinal disorders) | 1
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 1
HAEMATEMESIS (Gastrointestinal disorders) | 1
ILEUS (Gastrointestinal disorders) | 3
ILEUS PARALYTIC (Gastrointestinal disorders) | 2
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1
MELAENA (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2
STOMATITIS (Gastrointestinal disorders) | 2
SUBILEUS (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 6
CATHETER RELATED COMPLICATION (General disorders) | 4
CHEST PAIN (General disorders) | 4
CHILLS (General disorders) | 1
DEATH (General disorders) | 2
FATIGUE (General disorders) | 5
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 3
MUCOSAL INFLAMMATION (General disorders) | 2
MULTI-ORGAN FAILURE (General disorders) | 1
PYREXIA (General disorders) | 5
BILIARY DILATATION (Hepatobiliary disorders) | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1
CHOLESTASIS (Hepatobiliary disorders) | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 1
HEPATIC LESION (Hepatobiliary disorders) | 1
CATHETER RELATED INFECTION (Infections and infestations) | 4
ERYSIPELAS (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 2
HERPES SIMPLEX (Infections and infestations) | 1
INFECTION (Infections and infestations) | 1
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1
PARONYCHIA (Infections and infestations) | 2
PERITONEAL ABSCESS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 4
SEPSIS (Infections and infestations) | 1
SEPTIC SHOCK (Infections and infestations) | 1
SINUSITIS (Infections and infestations) | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 3
UROSEPSIS (Infections and infestations) | 2
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1
IATROGENIC INJURY (Injury, poisoning and procedural complications) | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1
WEIGHT DECREASED (Investigations) | 2
DEHYDRATION (Metabolism and nutrition disorders) | 5
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1
METABOLIC DISORDER (Metabolism and nutrition disorders) | 1
PODAGRA (Metabolism and nutrition disorders) | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1
BURSITIS (Musculoskeletal and connective tissue disorders) | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 1
COLORECTAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
HEMIPARESIS (Nervous system disorders) | 1
INTRACRANIAL VENOUS SINUS THROMBOSIS (Nervous system disorders) | 1
ISCHAEMIC STROKE (Nervous system disorders) | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1
VASCULITIS CEREBRAL (Nervous system disorders) | 1
HAEMATURIA (Renal and urinary disorders) | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 2
PYELOCALIECTASIS (Renal and urinary disorders) | 1
RENAL COLIC (Renal and urinary disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1
OVARIAN CYST (Reproductive system and breast disorders) | 1
PROSTATITIS (Reproductive system and breast disorders) | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2
LARYNGOSPASM (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 11
PULMONARY THROMBOSIS (Respiratory, thoracic and mediastinal disorders) | 1
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 2
CIRCULATORY COLLAPSE (Vascular disorders) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 4
HYPOTENSION (Vascular disorders) | 2
PHLEBITIS (Vascular disorders) | 1
THROMBOSIS (Vascular disorders) | 3
VENA CAVA THROMBOSIS (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus FOLFIRI (N=154)
ANAEMIA (Blood and lymphatic system disorders) | 18
LEUKOPENIA (Blood and lymphatic system disorders) | 8
NEUTROPENIA (Blood and lymphatic system disorders) | 50
VERTIGO (Ear and labyrinth disorders) | 13
CONJUNCTIVITIS (Eye disorders) | 33
DRY EYE (Eye disorders) | 10
LACRIMATION INCREASED (Eye disorders) | 8
ABDOMINAL PAIN (Gastrointestinal disorders) | 31
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 10
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 10
CONSTIPATION (Gastrointestinal disorders) | 46
DIARRHOEA (Gastrointestinal disorders) | 119
DYSPEPSIA (Gastrointestinal disorders) | 18
NAUSEA (Gastrointestinal disorders) | 85
STOMATITIS (Gastrointestinal disorders) | 39
VOMITING (Gastrointestinal disorders) | 41
ASTHENIA (General disorders) | 42
CHEST PAIN (General disorders) | 10
FATIGUE (General disorders) | 49
MUCOSAL INFLAMMATION (General disorders) | 40
OEDEMA PERIPHERAL (General disorders) | 18
PAIN (General disorders) | 10
PYREXIA (General disorders) | 19
NASOPHARYNGITIS (Infections and infestations) | 11
PARONYCHIA (Infections and infestations) | 37
RHINITIS (Infections and infestations) | 10
URINARY TRACT INFECTION (Infections and infestations) | 9
WEIGHT DECREASED (Investigations) | 21
ANOREXIA (Metabolism and nutrition disorders) | 34
HYPOKALAEMIA (Metabolism and nutrition disorders) | 35
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 29
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 9
DYSGEUSIA (Nervous system disorders) | 15
HEADACHE (Nervous system disorders) | 9
PARAESTHESIA (Nervous system disorders) | 9
POLYNEUROPATHY (Nervous system disorders) | 8
DEPRESSION (Psychiatric disorders) | 8
INSOMNIA (Psychiatric disorders) | 13
COUGH (Respiratory, thoracic and mediastinal disorders) | 12
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 16
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 18
ACNE (Skin and subcutaneous tissue disorders) | 55
ALOPECIA (Skin and subcutaneous tissue disorders) | 52
DERMATITIS (Skin and subcutaneous tissue disorders) | 9
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 32
DRY SKIN (Skin and subcutaneous tissue disorders) | 61
ERYTHEMA (Skin and subcutaneous tissue disorders) | 16
NAIL TOXICITY (Skin and subcutaneous tissue disorders) | 9
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 25
PRURITUS (Skin and subcutaneous tissue disorders) | 30
RASH (Skin and subcutaneous tissue disorders) | 64
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 31
SKIN TOXICITY (Skin and subcutaneous tissue disorders) | 18
HYPOTENSION (Vascular disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.